CLINICAL TRIAL: NCT03701438
Title: Immune Response to Influenza Vaccine in Subjects With B-cell Malignancies Treated With Idelalisib
Brief Title: Immune Response to Influenza Vaccine in Adults With B-cell Malignancies Treated With Idelalisib
Status: Terminated | Type: Observational
Why Stopped: The Swissmedic agency released Gilead from this post marketing requirement.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: GS-US-313-4100; 2017-003055-30 (EudraCT Number)
Record Dates: First submitted 2018-10-08; First posted 2018-10-10 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2019-11

CONDITIONS: B-cell Malignancies
MeSH Terms: interventions — Influenza Vaccines

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Idelalisib: Participants currently enrolled in a Gilead-sponsored study, who are currently being treated with 100 or 150 mg of idelalisib twice daily for at least 7 consecutive days prior to receiving an influenza vaccine.
  Interventions: Biological: Influenza Vaccine

INTERVENTIONS:
Biological: Influenza Vaccine — Administered per standard of care using a vaccine licensed and recommended in the site's country

SUMMARY:
The primary objective of this study is to assess the immune response to an influenza vaccine in adults with B-cell malignancies who are currently receiving treatment with idelalisib in a Gilead-sponsored study (parent study).

ELIGIBILITY:
Key Inclusion Criteria:

* Currently enrolled in a Gilead-sponsored study, receiving or scheduled to initiate treatment with idelalisib for at least 7 consecutive days prior to receiving an influenza vaccine
* Will be receiving an influenza vaccine per standard of care
* Willing to comply with scheduled visits, laboratory tests, other study procedures, and study restrictions
* Signed informed consent form, indicating that the subject has been informed of the procedures to be followed, potential risks and discomforts, and other pertinent aspects of study participation

Key Exclusion Criteria:

* Administration of systemic steroids for more than 2 consecutive weeks within the past 3 months (i.e., 12 weeks) prior to receiving an influenza vaccination. Up to 3 single doses of systemic corticosteroids (e.g., given as a premedication) are permitted within 30 days prior to receiving an influenza vaccine, however none of these doses may be administered within 7 days prior to influenza vaccination. Topical and inhaled steroids are permitted
* Intravenous immunoglobulin (IVIG) therapy within the past 3 months (i.e., 12 weeks) prior to receiving an influenza vaccination, and/or planned administration during the study period
* Cytotoxic chemotherapy and chronic administration (more than 14 days) of immunosuppressants within 30 days of vaccination
* Vaccination against influenza within the last 24 weeks prior to vaccination in this study, and/or planned administration of a second dose of influenza vaccine during the study period.
* Receipt of any vaccine in the 4 weeks preceding the trial vaccination or planned receipt of any vaccine in the 4 weeks following trial vaccination
* History of severe allergic or hypersensitivity reaction that is likely to be exacerbated by any component of an influenza vaccine including egg and chicken protein, or history of hypersensitivity to a previous dose of an influenza vaccine
* Acute disease and/or fever at the time of baseline blood draw (fever is defined as temperature ≥ 38°C in an oral setting)
* Presence of any condition that could, in the opinion of the investigator, compromise the subject's ability to participate in the study, such as history of substance abuse or psychiatric condition
* Females who are pregnant or lactating (refer to the Gilead-sponsored parent study's definition of 'child-bearing potential' to determine if pregnancy testing is required. If a pregnancy test has been performed in the Gilead-sponsored parent study ≤ 6 weeks prior to the baseline blood draw, it may be used for eligibility purposes.

Note: Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with B-cell malignancies currently receiving or initiating treatment with idelalisib in a Gilead-sponsored study.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2019-10-09 (Actual); Study Completion 2019-10-09 (Actual)

PRIMARY OUTCOMES:
Seroconversion Rate: Proportion of Participants with Either a Pre-Vaccination Hemagglutination Inhibition (HI) Titer < 1:10 and a Post-Vaccination HI titer ≥ 1:40, or a Pre-Vaccination HI titer ≥ 1:10 and a ≥ 4-fold Increase in Post-Vaccination HI Titer | 28 days [± 7 days] post-vaccination

SECONDARY OUTCOMES:
Seroprotection Rate: Proportion of Participants with HI titer ≥ 1:40 Post-Vaccination | 28 days [± 7 days] post-vaccination
Geometric Mean Titers (GMTs) of Antibodies: Pre- and Post-Vaccination GMTs of HI Antibodies Evaluated Prior to and 28 days (± 7 Days) After Vaccination | Prior to and 28 days (± 7 days) after vaccination
Percentage of Participants with Adverse Events or Serious Adverse Events From Time of Baseline Blood Draw Until Day 28 (Post Vaccination) Visit | Baseline Blood Draw; Day 28 (± 7 days)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (2):
- Fakultni nemocnice Kralovske Vinohrady, Interni hematologicka klinika, Prague, Czechia
- Hospital Universitario Ramon y Cajal, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy